CLINICAL TRIAL: NCT04689893
Title: Head-to-head Comparison of 68Ga-DOTA-TATE and 68Ga-DOTA-JR11 PET/CT in Patients With Tumor-induced Osteomalacia
Brief Title: Application of 68Ga-DOTA-TATE and 68Ga-DOTA-JR11 PET/CT in the Diagnosis and Evaluation of TIO
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PUMCHTIOJR11
Record Dates: First submitted 2020-12-28; First posted 2020-12-30 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Tumor-Induced Osteomalacia
MeSH Terms: conditions — Oncogenic osteomalacia | interventions — gallium Ga 68 dotatate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-DOTA-TATE and 68Ga-DOTA-JR11 PET/CT scan (Experimental): Patients of Tumor-induced osteomalacia PET/CT imaging: The patients were subcutaneously injected with 68Ga-DOTA-TATE and 68Ga-DOTA-JR11 and underwent PET/CT scan 20~40min after the injection in two consecutive days.
  Interventions: Drug: 68Ga-Dotatate; Drug: 68Ga-DOTA-JR11

INTERVENTIONS:
Drug: 68Ga-Dotatate — 68Ga-Dotatate was injected into the patients before the PET/CT scans
  Other Names: 68Ga-Dotatate injection
Drug: 68Ga-DOTA-JR11 — 68Ga-DOTA-JR11 was injected into the patients before the PET/CT scans
  Other Names: 68Ga-DOTA-JR11 injection

SUMMARY:
This is an open-label whole-body PET/CT study for investigating the value of 68Ga-DOTA-TATE and 68Ga-DOTA-JR11 PET/CT in patients with Tumor-induced osteomalacia.

DETAILED DESCRIPTION:
Tumor-induced osteomalacia (TIO), also known as oncogenic osteomalacia, is a rare paraneoplastic syndrome. The key to the cure of TIO is surgical resection of the culprit tumor. Over the last decade, 68Ga-labeled SSTR-based imaging has made a significant impact in detecting the culprit tumor of TIO 68Ga-DOTA-TATE is the most used SSTR PET tracer for the detection of TIO and it was recommended as first-line imaging method for localization of the causative tumor.

However, false positive, including fracture and/or inflammation, in 68Ga-DOTA-TATE PET/CT is a challenge in image interpretation, which may make the causative tumor indistinguishable in multiple suspicious lesions. There is no effective way to identify multiple suspicious lesions with intensive increased uptake on 68Ga-DOTA-TATE PET/CT.

68Ga-DOTA-JR11 is a SSTR2 specific antagonist used for PET tracer. However, the SSTR2 affinity of 68Ga-DOTA-JR11 is lower than 68Ga-DOTA-TATE, which means that the uptake of 68Ga-DOTA-JR11 by suspected lesions may be lower than that of 68Ga-DOTA-TATE. The purpose of this prospective study is to compare the sensitivity of 68Ga-DOTA-JR11 and 68Ga-DOTA-TATE PET/CT for detecting the responsible tumor of TIO and investigate if 68Ga-DOTA-JR11 PET/CT can identify the culprit tumor of TIO in multiple suspicious lesions.

ELIGIBILITY:
Inclusion Criteria:

* suspected or confirmed untreated TIO patients;
* 68Ga-DOTA-TATE and 68Ga-DOTA-JR11 PET/CT within two weeks;
* signed written consent.

Exclusion Criteria:

* pregnancy;
* breastfeeding;
* any medical condition that in the opinion of the investigator may significantly interfere with study compliance.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-03-15 (Actual); Primary Completion 2021-03-15 (Estimated); Study Completion 2022-03-15 (Estimated)

PRIMARY OUTCOMES:
Diagnostic value | through study completion, an average of 1 year
  Sensitivity and Specificity of 68Ga-DOTA-JR11 PET/CT for TIO in comparison with 68Ga-DOTATATE PET/CT

CONTACTS AND LOCATIONS:
Overall Officials: Hongli Jing, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking union medical college hospital, Beijing, Dongcheng, China

REFERENCES:
- [Derived] Hou G, Zhang Y, Liu Y, Wang P, Xia W, Xing X, Huo L, Li F, Jing H. Head-to-Head Comparison of 68Ga-DOTA-TATE and 68Ga-DOTA-JR11 PET/CT in Patients With Tumor-Induced Osteomalacia: A Prospective Study. Front Oncol. 2022 Feb 24;12:811209. doi: 10.3389/fonc.2022.811209. eCollection 2022. PMID 35280786